CLINICAL TRIAL: NCT03978533
Title: Low Intensity Family Support for Refugees in an LMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stevan Weine, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0547; R21MH117759 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-06-07 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Depression; Anxiety; PTSD; Family Dynamics
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Support Group (Experimental): Family Support Groups will be piloted with families in community and clinical sites. Each pair of facilitators will pilot two groups of 6 families each. Each group is 4 sessions lasting 2 hours each. Each of the sessions incorporates didactic talks, family discussion, and separate breakout groups for adolescents and adults. Family Support intervention incorporates cognitive-behavioral theory of PM+ which underlies evidence-based techniques focused on stress management and behavioral activation. Family support intervention also incorporates resilience theory, which explains family protective processes that can ameliorate the negative consequences of hardships and challenges and enable healing and growth in families.
  Interventions: Behavioral: Family Support Group

INTERVENTIONS:
Behavioral: Family Support Group — Family Support Groups will be piloted with families in community and clinical sites. Each pair of facilitators will pilot two groups of 6 families each. Each group is 4 sessions lasting 2 hours each. Each of the sessions incorporates didactic talks, family discussion, and separate breakout groups for adolescents and adults. Family Support intervention incorporates cognitive-behavioral theory of PM+ which underlies evidence-based techniques focused on stress management and behavioral activation. Family support intervention also incorporates resilience theory, which explains family protective processes that can ameliorate the negative consequences of hardships and challenges and enable healing and growth in families.

SUMMARY:
The rapidly growing scale of humanitarian crises requires new response capabilities geared towards addressing populations with prolonged high vulnerability to mental health consequences and little to no access to mental health, health, and social resources. This R21 develops and pilot tests a novel model for helping urban refugee families in LMICs with little to no access to evidence-based mental health services, by delivering a transdiagnostic family intervention for common mental disorders in health sector and non-health sector settings. The project is located in Istanbul, Turkey. Aim 1 forms a Family Support Design Team (FSDT) to adopt the PM+ and CAFES manuals into a family support (FS) intervention for use with refugee families by lay providers in community sites and nurses in clinical sites using a four-session multiple family group format. Aim 2 pilots FS with families in community and clinical sites, and then through observations and qualitative interviews, assesses FS's feasibility, fidelity, the impact of context and local capacity, the experiences of intervention delivery, and practitioner and organizational perspectives on scale up. Aim 3 conducts pre, immediate post, and 3-month post assessments of the refugee families who received FS through all the sites, to demonstrate the kind of pre-post changes that have been reported for comparable interventions and to determine key parameters of interest with sufficient accuracy and precision. This exploratory investigation, conducted with the support and advice of the World Health Organization, will strengthen the research capabilities of the academic and community partners in Istanbul and will develop new evidence-based mental health services for refugees in Turkey and other LMICs, as well as for refugees and migrants in low resource communities in the United States.

DETAILED DESCRIPTION:
RATIONALE The rapidly growing scale of global humanitarian crises requires new response capabilities geared towards addressing populations with prolonged high vulnerability to mental health consequences and little access to health and social resources. The World Health Organization (WHO), under the leadership of Dr. Mark van Ommeren, has been advocating for low resource-intensity cognitive behavioral therapy (LICBT) for such conditions. They conducted two large RCTs of Problem Management Plus (PM+), a brief, basic, one-on-one, paraprofessional-delivered version of LICBT for adults, which demonstrated clinically significant reductions in anxiety and depressive symptoms at 3 months. LICBT could help to address some needs among Syrian refugees, but our recent D43 supported longitudinal study of 30 Syrian refugee families in Istanbul, found that one key challenge is its fit with the strong family context of Syrians. The investigators found evidence of families with adult and/or children with CMD symptoms and challenges managing stress, but also evidence of family strengths and resilience, and families facing multiple adverse challenges. In August 2017, Dr. Weine met with Dr. van Ommeren at the WHO, and they agreed to work in partnership to extend the WHO's LICBT approach to families. In September 2017, Weine et al convened a roundtable with key stakeholders in Istanbul, which reached a consensus about the need for a new family intervention that included elements of PM+ but also of family interventions, for delivery in a group format. Specifically, the investigators chose to incorporate elements of Coffee and Families Education and Support (CAFES), a NIMH funded family support and education intervention that the investigators previously developed and evaluated with refugee families from Bosnia and Kosovo. Other key implementation challenges are who will conduct the intervention, what training do they require, what organizational capacity is required, and how to best integrate FS into community and clinical sites.

AIM 1 To form a Family Support Design Team (FSDT) to adopt the PM+ and CAFES manuals into a family support (FS) intervention for use with Syrian refugee families by lay providers in community sites and nurses in clinical sites using a four-session multiple family group format.

AIM 2 To pilot FS with families in community and clinical sites, and then through observations and qualitative interviews, to assess FS's feasibility, fidelity, the impact of context and local capacity, the experiences of intervention delivery, and practitioner and organizational perspectives on scale up.

AIM 3 To conduct pre, immediate post, and 3-month post assessments of the Syrian refugee families who received FS through all the sites, to demonstrate the kind of pre-post changes that have been reported for comparable interventions and to determine key parameters of interest with sufficient accuracy and precision.

ELIGIBILITY:
Inclusion Criteria:

* Syrian refugee family living in Istanbul
* contains both adult caregivers (18-55) and at least one of their children (<18 and >11 years) living in one household
* one adult or adolescent with > 3 on the GHQ-12
* willing to participate in the intervention and research procedures
* able to give written informed consent

Exclusion Criteria:

• Families who do no have a child <18 and >11 years old

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 189 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Strengths and Difficulties Questionnaire at immediate post and three months post intervention | baseline, immediate post, three months post
  Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire about 3-16 year olds. For this project, the adolescent version will be used for ages 11-17. The questionnaire comprises 5 scales of 5 items each. Total difficulties score: This is generated by summing scores from all the scales except the prosocial scale.
  Scoring is close to average; slightly raised (/slightly lowered); high (/low); very high (very low)
  Total difficulties score: 0-14; 15-17; 18-19; 20-40
  Emotional problems score: 0-4; 5; 6; 7-10
  Conduct problems score: 0-3; 4; 5; 6-10
  Hyperactivity score: 0-5; 6; 7; 8-10
  Peer problems score: 0-2; 3; 4; 5-10
  Prosocial score:7-10; 6; 5; 0-4
Change from baseline of Kansas Parental Satisfaction Scale at immediate post and three months post intervention | baseline, immediate post, three months post
  Kansas Parental Satisfaction Scale (KPSS) asks three questions about their satisfaction with a) their children's behavior, b) them as a parent, and c) their relationship with their children. The instrument uses a 7-point Likert scale with response choices ranging from 1 ("extremely dissatisfied") to 7 ("extremely satisfied"). The scores for all three items are summed to yield a total parenting satisfaction score. Scores range from 3 - 21. Scores of 15 or less indicate low parental satisfaction.
Change from baseline of PTSD Checklist for DSM-5 at immediate post and three months post intervention | baseline, immediate post, three months post
  PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including: Monitoring symptom change during and after treatment; Screening individuals for PTSD; Making a provisional PTSD diagnosis. The PCL-5 is a self-report measure that can be completed by patients in a waiting room prior to a session or by participants as part of a research study. It takes approximately 5-10 minutes to complete.The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." Treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 Criterion B item (questions 1-5), 1 Criterion C item (questions 6-7), 2 Criterion D items (questions 8-14), 2 Criterion E items (questions 15-20).
Change from baseline Hospital Anxiety Depression Scale at immediate post and three months post intervention | baseline, immediate post, three months post
  HADS (Hospital Anxiety and Depression Scale) aims to measure symptoms of anxiety (HADS Anxiety) and depression (HADS Depression).The HADS is a fourteen item scale; seven of the items relate to anxiety and seven relate to depression. Each question is scored 0-3, a person can score between 0 and 21 for either anxiety or depression. For both scales of depression or anxiety, a score of 0-7 is normal, 8-10 is mild, 11-14 is moderate, and 15-21 is severe.
Change from baseline General Health Questionnaire at immediate post and three month post intervention | baseline, immediate post, three months post
  General Health Questionnaire (GHQ-12) is a screening device for identifying minor psychiatric disorders in the general population. The GHQ-12 is a quick, reliable and sensitive short form that is ideal for research studies. The GHQ-12 yields an overall total score. The GHQ scoring is 0-0-1-1, with a score range from 0-12. Any score exceeding the threshold value of 3 as achieving 'caseness'.

SECONDARY OUTCOMES:
Change from baseline Family Communication Questionnaire at immediate post and three month post intervention | baseline, immediate post, three months post
  Family Communication Questionnaire is a measure that assess how often and how comfortable the family is about communicating on certain issues. There are six items, each with a question on how often they talk about an issue (responses include: a lot, often, once in a while, we don't talk about this) and a question on how comfortable they are talking about the issue asked (responses include: very comfortable, somewhat comfortable, somewhat uncomfortable, very very uncomfortable) for a total of 12 items that are scored 0-3, for a total score of 36. High scores indicate low family communication, with cut of score of 24 and above for low family communication.
Change in baseline Knowledge and Attitudes Regarding Trauma Mental Health Questionnaire at immediate post and three month post intervention | baseline, immediate post, three months post
  This construct is assessed using a 28 item questionnaire. There are two sub-scales that assess knowledge and attitude. The knowledge sub-scale (13 items) presents items with varying level of difficulty to address the degree to which the subject is informed about the conditions and treatment of PTSD and Depression, and cost, availability, and accessibility of services. Items are scored for "true," "false," or "can't say". There is no total score, rather assessing their change in knowledge over time.
  The attitude sub-scale (15 items) assesses the degree to which subjects consider the trauma related mental health problems to be addressable. Items are scored on a 4-point scale from 0-4 for "strongly agree" to "strongly disagree" for a total score of 60. Some items are reverse scored, a score of 30 or higher indicates positive attitudes and below 30 indicates negative attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Stevan Weine, MD, Principal Investigator — University of Illinois at Chicago
Locations (6):
- Turkey (Türkiye) (6):
  - Can Association, Istanbul
  - Hiraeth, Istanbul
  - Insan for Psychosocial Support, Istanbul
  - Syrian Nour Association, Istanbul
  - Turkish Red Crescent, Istanbul
  - Yusra Community Center, Istanbul

IPD SHARING:
Plan to Share IPD: No